CLINICAL TRIAL: NCT02968069
Title: Development and Validation of a Predictive Model for Early Gastric Cancerous Lesions Under Endoscopic Observation
Brief Title: A Predictive Model Based on Narrow Band Imaging for Early Gastric Cancerous Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Putuo District Center Hospital (Other); Shanghai MCC worker hospital (Unknown)
Responsible Party: Principal Investigator, Xiaobo Li, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-138k
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected gastric cancerous lesions (Experimental): Magnifying endoscopy with NBI would be conducted for every patient included in our study
  Interventions: Device: NBI

INTERVENTIONS:
Device: NBI — Endoscopic factors under white light view and simplified narrow band imaging classification assisting in diagnosing cancerous lesions will be recorded.
  Other Names: Evis Lucera system (CV-260, Olympus Inc, Japan); high-definition colonoscopes (CF-H260AL, Olympus Inc, Japan); magnifying colonoscopes (CF-H260AZL, Olympus Inc, Japan)

SUMMARY:
Without high diagnostic efficacy of endoscopic forceps biopsy (EFB) and with low diagnostic efficacy of narrow band imaging (NBI) in novice endoscopists and endoscopists of community hospitals in China, it is urgent to improve diagnostic efficacy for gastric cancerous lesions.The investigators will conduct a study to develop and validate a diagnostic model based on NBI for early gastric cancerous lesions under endoscopic observation.

DETAILED DESCRIPTION:
Endoscopic forceps biopsy (EFB) is considered the gold standard and most commonly used for histological diagnosis of gastric epithelial neoplasia before proper management.Many studies have shown that there exist considerable discrepancies between EFB and subsequently resected specimens with discrepancy rate of 27.1-44.5%. On the other hand, with low diagnostic efficacy of narrow band imaging (NBI) in novice endoscopists and endoscopists of community hospitals in China, not higher diagnostic accuracy of gastric cancerous lesions could be observed. Here, the investigators will conduct a study to develop and validate a diagnostic model based on narrow band imaging for early gastric cancerous lesions under endoscopic observation, trying to improve overall diagnostic efficacy for gastric cancerous lesions.

ELIGIBILITY:
Inclusion Criteria:

* Suspected of having a cancerous lesions
* The age of patients is from 40-80 years
* Patients must undergo esophagogastroduodenoscopy

Exclusion Criteria:

* Clinical diagnosis of advanced gastric cancer
* Acute upper gastrointestinal bleeding
* Severe systemic diseases
* Refuse to attend the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the diagnostic model in histological prediction of gastric cancerous lesions | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Li, MD.Ph.D, Principal Investigator — Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai,China,Shanghai Institute of Digestive Disease, Shanghai

IPD SHARING:
Plan to Share IPD: No